CLINICAL TRIAL: NCT04727957
Title: Predictive Analytics in Ventilator-Associated Events
Brief Title: Predictive Analytics in Lower Respiratory Tract Infections (VA-LRTIs)
Acronym: PA in VA-LRTIs
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Miia M Jansson, PhD, Adjunct Professor, PhD, University of Oulu
Other Study IDs: University of Oulu
Record Dates: First submitted 2021-01-05; First posted 2021-01-27 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Ventilator-Associated Event

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dataset for development and testing
  Interventions: Other: Diagnostic and prognostic models for VA-LRTIs
- Dataset for external validation
  Interventions: Other: Diagnostic and prognostic models for VA-LRTIs

INTERVENTIONS:
Other: Diagnostic and prognostic models for VA-LRTIs — Diagnostic and prognostic models for VA-LRTIs

SUMMARY:
To determine the accuracy and generalizability of VA-LRTI algorithm to detect and predict three high-incidence and high-impact VAEs from electronic health records data: 1) ventilator-associated event, 2) ventilator-associated pneumonia, and 3) ventilator-associated tracheobronchitis.

ELIGIBILITY:
All invasively ventilated ICU patient (aged 18 or over)

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adult mixed medical-surgical ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with VA-LRTI as assessed by risk-calculator | 1.6.-31.12.2021
  Prediction model to be used at the moment of diagnosis and algorithms to be used prior IMV to predict the risk of VA-LRTI.

SECONDARY OUTCOMES:
Rate of in-hospital mortality | 1.6.-31.12.2021
  Prediction model to be used at the moment of diagnosis to predict the risk of mortality in VA-LRTIs.

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy of Oulu, Oulu, Finland

IPD SHARING:
Plan to Share IPD: Undecided